CLINICAL TRIAL: NCT05326490
Title: A Multi-center, Randomized, Double-Blinded, Parallel and Placebo-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of PB-201 in Type 2 Diabetic Mellitus Patients With Poor Glycemic Control Via Metformin Hydrochloride Monotherapy
Brief Title: Study to Evaluate the Efficacy and Safety of PB-201 in Type 2 Diabetic Mellitus Patients With Poor Glycemic Control Via Metformin Hydrochloride Monotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB201302
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Lead-201; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test arm (Experimental): Double-blinded treatment period:
  PB201 100 mg, one tablet in the morning and one tablet in the evening;Basic treatment with stable dose of Glucophage
  Open-label extended period:
  PB201 100 mg, one tablet in the morning and one tablet in the evening;Basic treatment with stable dose of Glucophage
  Interventions: Drug: PB-201; Drug: Metformin hydrochloride
- Placebo arm (Placebo Comparator): Double-blinded treatment period:
  PB-201 matched placebo: One tablet each time, orally in the morning and evening respectively;Basic treatment with stable dose of Glucophage
  Open-label extended period:
  PB201 100 mg, one tablet in the morning and one tablet in the evening;Basic treatment with stable dose of Glucophage
  Interventions: Drug: PB-201 matched placebo; Drug: Metformin hydrochloride

INTERVENTIONS:
Drug: PB-201 — PB-201: 100 mg each time, orally in the morning and evening respectively
  Arms: Test arm
Drug: PB-201 matched placebo — PB-201 matched placebo: One tablet each time, orally in the morning and evening respectively
  Arms: Placebo arm
Drug: Metformin hydrochloride — The dosage and administration of metformin hydrochloride remain unchanged before screening

SUMMARY:
This is a Multi-center, Randomized, Double-Blinded, Parallel and Placebo-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of PB-201 in Type 2 Diabetic Mellitus Patients with Poor Glycemic Control via Metformin Hydrochloride Monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for this study:

  1. Males or females aged ≥18 years and ≤ 75 years at screening;
  2. Definitely diagnosed T2DM patients who meet the diagnostic criteria for type 2 diabetes mellitus issued by WHO in 1999;
  3. Receive a stable dose of metformin hydrochloride monotherapy ≥ 8 weeks on the basis of diet and exercise interventions before screening and the dose of metformin hydrochloride is ≥ 1500mg/day or the maximum tolerated dose (<1500mg/day but ≥ 1000mg/day);
  4. The Glycosylated hemoglobin (HbA1c) must meet the following criteria:

     HbA1c ≥ 7.5% and ≤ 11.0% at screening (local laboratory); HbA1c ≥ 7.0% and ≤ 10.5% (central laboratory) prior to randomization(V3);
  5. Fasting plasma glucose (FPG) must meet the following criteria:

     FPG < 15 mmol/l at screening (local laboratory); FPG < 15 mmol/l (central laboratory) prior to randomization (V3);
  6. Body mass index (BMI) ≥ 18.5 kg/m2 and ≤ 40.0 kg/m2 at screening or prior to randomization (V3);
  7. Able to understand and willing to sign the written informed consent form (ICF) and follow the protocol.

Exclusion Criteria:

* Patients cannot be randomized if they meet any of the following criteria:

  1. Patients diagnosed with type 1 diabetes mellitus, diabetes due to pancreatic injury, or special type of diabetes due to other diseases (e.g., acromegaly or Cushing's syndrome);
  2. Fasting C-peptide < 0.8 ng/mL at screening;
  3. Patients who use other hypoglycemic drugs except metformin, systemic glucocorticoids (except inhalation or topical external use) and growth hormones within eight weeks before screening or prior to randomization;
  4. Patients who use insulin continuously for more than 14 days within six months before screening or prior to randomization (the time of insulin treatment for gestational diabetes mellitus is not within this limit);
  5. Patients who receive other glucokinase activators prior to screening or randomization;
  6. Patients who have acute diabetic complications such as diabetic ketoacidosis, lactic acidosis or hyperglycemia and hyperglycemic hyperosmolar status within six months before screening or prior to randomization;
  7. Patients who have severe chronic diabetic complications (such as proliferative diabetic retinopathy, severe diabetic neuropathy, diabetic foot, etc.) within six months before screening.
  8. Patients who have two or more episodes of severe hypoglycemia within sixmonths before screening, or who have had severe hypoglycemia prior to randomization since screening;
  9. Patients who develop any of the following heart diseases within six months before screening or prior to randomization:

     Decompensated cardiac insufficiency (New York Heart Association NYHA Classification of grade III or IV); Acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting, or coronary artery balloon dilates or coronary stent implantation; Severe arrhythmias (e.g., second- or third-degree atrioventricular block, long QT syndrome, or QTcF > 480 ms); Arrhythmias that require treatment, or other arrhythmias assessed by the investigator as unsuitable for participation in this clinical study;
  10. Patients whose hypertension symptoms are not effectively controlled at screening or prior to randomization (sitting systolic blood pressure ≥160mmHg and/or sitting diastolic blood pressure ≥ 100mmHg after resting ≥5 minutes);
  11. Patients who have hemorrhagic stroke or acute ischemic stroke within six months before screening or prior to randomization;
  12. Patients who have severe kidney disease or estimated glomerular filtration rate eGFR < 60mL/(min 1.73 m2) or in routine urine qualitative proteinuria ≥ (++) or quantitative proteinuria ≥1 g/L at screening or prior to randomization;
  13. Patients who have a history of acute or chronic pancreatitis at screening or prior to randomization;
  14. Patients who suffer from any serious gastrointestinal diseases (such as gastroparesis, inflammatory bowel disease, intestinal obstruction) that affect drug absorption within six months before screening or prior to randomization,or undergo gastrointestinal operations that affect drug absorption (such as gastrectomy, gastroenterostomy or enterectomy, etc.);
  15. Patients who have severe trauma or serious infection that may affect glycaemic control within one month before screening or prior to randomization, such as fracture, pneumonia, etc.;
  16. Patients with any type of treated or untreated malignancy (whether cured or not) within five years before screening or prior to randomization. However,patients with cured basal cell carcinoma of the skin do not need to be excluded;
  17. Patients with thyroid dysfunction not controlled by stable drug dosage at screening or with clinically significant thyroid function test abnormalities at screening and requiring medical treatment;
  18. Patients who have any of the following laboratory abnormalities at screening:

      Human immunodeficiency virus antibody or Treponema pallidum specific antibody positive; Hepatitis C antibody positive; Hepatitis B surface antigen is positive, and the result of hepatitis B virus DNA quantitative test is higher than the lower limit of the test reference range (Note: If the local laboratory cannot carry out quantitative detection of hepatitis B virus, the sample will be sent to the central laboratory.);
  19. Patients who have any of the following laboratory abnormalities at screening or prior to randomization:

      Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN), or total bilirubin > 1.5×ULN; Hemoglobin < 110 g/L; Fasting triglycerides ≥ 5.7 mmol/L;
  20. Patients who have any disease at screening or prior to randomization that may cause hemolysis or red blood cell instability affecting HbA1c testing, such as hemolytic anemia;
  21. Patients who have a history of blood donation, transfusion, or loss of > 400 ml within ninety days before screening or prior to randomization;
  22. Subject who has participated in any drug or medical device clinical study within three months before screening or prior to randomization (except those who fail in screening or do not receive any test drug);
  23. Patients who have a prior history of clearly diagnosed psychiatric disorders, unwilling or unable to fully understand and cooperate, or assessed by the investigator as unsuitable for participation in this clinical study;
  24. Patients who have a prior history of drinking [(>2 units of alcohol per day and >14 units of alcohol per week (one unit of alcohol corresponds to 150mL of wine or 350mL of beer or 50 mL of spirits)] or history of drug abuse;
  25. Patients who are known to be allergic or intolerant to the test drug or Vildagliptin or its excipients, or who have contraindications;
  26. Patients who are currently being treated with strong or moderate liver enzyme CYP3A4 inducers;
  27. Female in pregnancy or lactation period;
  28. Partners of male subjects or female subjects who plan to become pregnant or who are unable or unwilling to use contraceptive methods approved by the protocol from the signing of the informed consent form to 30 days after the last use of the drug;
  29. Compliance with metformin or placebo < 80% or > 120% during single-blind run-in period;
  30. The investigator judges that the subject is unable to comply with the protocol requirements, such as unable to adhere to diet and exercise treatment during the study, unable to take drugs and meals on time according to the protocol requirements, and unable to conduct self-monitoring of blood glucose (SMBG) in time and record;
  31. Other circumstances that, in the opinion of the investigator, are not appropriate for participation in this clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2024-09-24 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Week 1,Week 25
  Change of glycosylated hemoglobin (HbA1c) from baseline to 24 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No